CLINICAL TRIAL: NCT01294293
Title: A Phase I Study of VTX-2337 in Combination With Pegylated Liposomal Doxorubicin (PLD; NSC# 712227) or in Combination With Weekly Pactilaxel (NSC #673089) in Patients With Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: TLR8 Agonist VTX-2337 and Pegylated Liposomal Doxorubicin Hydrochloride or Paclitaxel in Treating Patients With Recurrent or Persistent Ovarian Epithelial, Fallopian Tube, or Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9925; NCI-2011-02663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000695034; GOG-9925 (Other: NRG Oncology); GOG-9925 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Malignant Ovarian Mixed Epithelial Tumor; Ovarian Brenner Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — VTX-2337; Paclitaxel; Taxes

ARMS (1):
- Treatment (TLR8 agonist VTX-2337, PLD, and Paclitaxel) (Experimental): Patients receive TLR8 agonist VTX-2337 SC on days 3, 10, and 17 and pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 or TLR8 agonist VTX-2337 SC on days 1, 8, and 15 and paclitaxel IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: TLR8 Agonist VTX-2337; Other: Diagnostic Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Drug: Paclitaxel

INTERVENTIONS:
Drug: TLR8 Agonist VTX-2337 — Given SC
  Other Names: Toll-like Receptor 8 Agonist VTX-2337; VTX-2337
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: doxorubicin HCl liposome; TLC D-99
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; TAX

SUMMARY:
This phase I trial is studying the side effects and best dose of TLR8 agonist VTX-2337 and pegylated liposomal doxorubicin hydrochloride in treating patients with recurrent or persistent ovarian epithelial, fallopian tube, or peritoneal cavity cancer. Biological therapies, such as TLR8 agonist VTX-2337, may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as pegylated liposomal doxorubicin hydrochloride and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving TLR8 agonist VTX-2337 together with pegylated liposomal doxorubicin hydrochloride or paclitaxel may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated doses (MTD) and dose limiting toxicities (DLTs) of VTX-2337 when administered in combination with pegylated liposomal doxorubicin (PLD; Doxil, Lipodox™) 40 mg/m2 in Regimen 1 and when administered in combination with weekly paclitaxel 80 mg/m2 in Regimen 2, and the associated DLTs based on adverse events that occur in cycle 1 for each of these combinations in women with recurrent or persistent, epithelial ovarian, fallopian tube or primary peritoneal cancer.

II. To examine the tolerability of the combination at the MTD of VTX-2337 assessed in combination with PLD 40 mg/m2 and with PLD 50 mg/m2 in Regimen 1 and in combination with weekly paclitaxel in Regimen 2.

III. To determine recommended phase II doses (RP2D) of VTX-2337 in combination with PLD in Regimen 1 and in combination with weekly paclitaxel in Regimen 2.

SECONDARY OBJECTIVES:

I. To assess the biological effects (immune activation) of VTX-2337 in combination with PLD in Regimen 1 and in combination with weekly paclitaxel in Regimen 2.

II. To assess the pharmacokinetics in patients receiving VTX-2337 in combination with PLD in Regimen 1 and in combination with weekly paclitaxel in Regimen 2.

III. To assess the tolerability (including CTCAE v4 Grade 3/4 allergic reaction) of weekly paclitaxel 80 mg/m2 when administered without corticosteroid premedication (Regimen 2 only).

TERTIARY OBJECTIVES:

I. To assess the anti-tumor activity of VTX-2337 when administered concomitantly with PLD in Regimen 1 and when administered concomitantly with weekly paclitaxel in Regimen 2 in patients with recurrent or persistent epithelial ovarian fallopian tube or primary peritoneal cancer.

II. To assess the effect of TLR8 polymorphisms on the biological (immune) and clinical effects of VTX-2337 in combination with PLD in Regimen 1 and in combination with weekly paclitaxel in Regimen 2.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive TLR8 agonist VTX-2337 subcutaneously (SC) on days 3, 10, and 17 and pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 or TLR8 agonist VTX-2337 subcutaneously on days 1, 8, and 15 and paclitaxel IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically during courses 1 and 2 for pharmacokinetic, pharmacogenomic, and other research studies. After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma

  * Histologic documentation of the original primary tumor is required via the pathology report
* Patients with the following histologic cell types are eligible:

  * Serous adenocarcinoma
  * Endometrioid adenocarcinoma
  * Mucinous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial adenocarcinoma
  * Transitional cell carcinoma
  * Malignant Brenner tumor
  * Adenocarcinoma not otherwise specified (N.O.S.)
* Patient must have measurable disease or detectable (non-measurable) disease:

  * Measurable disease will be defined by RECIST 1.1

    * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded)
    * Each lesion must be ≥ 10 mm when measured by CT, MRI, or caliper measurement by clinical exam or ≥ 20 mm when measured by chest x-ray
    * Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI
  * Detectable (non-measurable) disease is defined as not having measurable disease but has at least one of the following conditions:

    * Baseline values of CA-125 ≥ 2 x ULN

      * Patients whose CA-125 is < 100 U/mL must undergo a second confirmatory value within a period of ≤ 4 weeks
      * Patients with a level ≥ 100 U/mL may be entered without confirmatory measurement
      * The CA-125 assessment for eligibility must be done at least 4 weeks after paracentesis or other surgical procedures
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions
  * Patient with measurable disease must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1

    * Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment

  * For patients enrolled in Regimen 2, weekly paclitaxel, treatment for their primary disease must have included paclitaxel; this can have been given weekly or every 3 weeks; patients who experienced severe hypersensitivity to paclitaxel are excluded
  * Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen

    * For patients enrolled in Regimen 1 which includes PLD, prior treatment with PLD is NOT allowed
    * For patients enrolled in Regimen 2 which includes weekly paclitaxel, prior treatment with weekly paclitaxel for recurrent or persistent disease is NOT allowed
  * Patients are allowed to receive, but are not required to receive, non-cytotoxic therapy (such as bevacizumab) as part of their primary treatment regimen; patients are allowed to receive, but are not required to receive, non-cytotoxic therapy for management of recurrent or persistent disease
  * Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* No patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA), or subarachnoid hemorrhage within six months of the first date of treatment on this study
* No patients who have received oral or parenteral corticosteroids within 2 weeks of study entry or who require ongoing systemic immunosuppressive therapy for any reason
* Patients must have a GOG performance status of 0 or 1
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3; this ANC cannot have been induced or supported by granulocyte colony-stimulating factors
* Platelets ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 x institutional upper limit normal (ULN)
* Bilirubin ≤ 1.5 x ULN
* SGOT (AST) ≤ 3.0 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Neuropathy (sensory and motor) less than or equal to grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Patients of childbearing potential must be practicing an effective form of contraception
* Patients should be free of active infection requiring parenteral antibiotics
* No patients with active autoimmune disease

  * "Active" refers to any condition currently requiring therapy
  * Examples of autoimmune disease include systemic lupus erythematosus, multiple sclerosis, inflammatory bowel disease, and rheumatoid arthritis
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer or localized cancer of the breast, head and neck, or skin, are excluded if there is any evidence of other malignancy being present within the last three years
* No patients with known chronic or active hepatitis
* No patients with clinically significant cardiovascular disease, this includes:

  * Uncontrolled hypertension, defined as systolic > 140 mm Hg or diastolic > 90 mm Hg
  * Myocardial infarction or unstable angina within 6 months of the first date of treatment on this study
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
  * QTc interval ≥ 450 ms on baseline ECG
  * Baseline ejection fraction ≤ 50% as assessed by echocardiogram or MUGA
  * New York Heart Association (NYHA) class II or higher congestive heart failure
  * Grade 2 or higher peripheral ischemia (brief [< 24 hours] episode of ischemia managed non-surgically and without permanent deficit)
* No patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration or nutrition
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration

  * Continuation of hormone replacement therapy is permitted
* No patients who have had previous treatment with VTX-2337, pegylated liposomal doxorubicin, doxorubicin, or any other anthracycline
* Patients are excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen (prior treatment with pegylated liposomal doxorubicin is NOT allowed)
* Patients are allowed to receive, but are not required to receive, non-cytotoxic therapy (such as bevacizumab) as part of their primary treatment regimen
* Patients are allowed to receive, but are not required to receive, non-cytotoxic therapy for management of recurrent or persistent disease
* Patients must have recovered from effects of recent surgery, radiotherapy, or chemotherapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded

  * Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube or primary peritoneal cancer within the last three years are excluded

  * Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* No patients who have received an investigational agent within 30 days of study entry
* Any other prior therapy directed at the malignant tumor, including biological and immunologic agents, must be discontinued at least three weeks prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
First-cycle dose-limiting toxicities | 28 days
Frequency and severity of toxicities as assessed by CTCAE | Up to 1 year

SECONDARY OUTCOMES:
Immune activation (e.g., Th1, cytokines) | Up to 1 year
  Immune response endpoints (e.g., Th1 cytokines) will be summarized with simple descriptive statistics and analyzed with linear mixed models accounting for the longitudinal aspect of the data.
Pharmacokinetic measures of TLR8 agonist VTX-2337 | Baseline, 0.5, 2, 4, 8, and 24 hours after TLR8 agonist VTX-2337 injection
Pharmacokinetic measures of pegylated liposomal doxorubicin hydrochloride | Baseline, 0.5, 2, 4, 8, and 24 hours after TLR8 agonist VTX-2337 injection
Pharmacokinetic measures of paclitaxel | Baseline, 0.5, 2, 4, 8, and 24 hours after TLR8 agonist VTX-2337 injection

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Monk, Principal Investigator — NRG Oncology
Locations (10):
- United States (10):
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island